CLINICAL TRIAL: NCT05589597
Title: A Global Multicenter Phase 1/2 Trial of EO4010, a Novel Microbial Derived Peptide Therapeutic Vaccine, in Combination With Nivolumab and/or Bevacizumab, for Treatment of Patients With Previously Treated Metastatic Colorectal Carcinoma
Brief Title: EO4010 in Previously Treated Metastatic Colorectal Carcinoma
Acronym: AUDREY
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to stop recruitment in context of overall EO4010 development goals. Stop of recruitment was not related to any safety concern, with the safety profile of EO4010 being benign
Sponsor: Enterome (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EOCRC2-22
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Nivolumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Multi-cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): E04010 Monotherapy
  Interventions: Drug: EO4010
- Cohort 2 (Experimental): E04010 in combination with nivolumab
  Interventions: Drug: EO4010
- Cohort 3 (Experimental): E04010 in combination with nivolumab and/or bevacizumab
  Interventions: Drug: EO4010

INTERVENTIONS:
Drug: EO4010 — Sequential assignment
  Other Names: Nivolumab; Bevacizumab

SUMMARY:
Open-label multicenter study

DETAILED DESCRIPTION:
This is an open-label, multicenter, FIH, phase 1/2 trial to assess safety, tolerability, immunogenicity, and preliminary efficacy of the microbial-derived therapeutic vaccine EO4010 in combination with nivolumab and/or bevacizumab for treatment of patients with unresectable, previously treated, metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent
2. Histological confirmation of advanced non-resectable colorectal adenocarcinoma
3. Patients with metastatic colorectal cancer who have been previously treated with, or are not considered candidates for
4. Progression during or within 3 months following the latest administration of standard therapies
5. Age ≥ 18 years old
6. Human leukocyte antigen (HLA)-A2 positive
7. ECOG performance status 0 or 1
8. Measurable disease according to Response Evaluation Criteria in Solid Tumors criteria (RECIST)
9. Patients with a life expectancy of at least 3 months
10. Female patients of childbearing potential must have a negative serum pregnancy test
11. Patients following recommendations for contraception
12. Patients willing and able to comply with the study procedures

Exclusion Criteria:

1. Patients treated with dexamethasone > 2 mg/day or equivalent within 14 days before randomization, unless required to treat an adverse event
2. Patients treated with radiotherapy within 12 weeks, and cytotoxic chemotherapy therapy within 28 days
3. Patients with persistent Grade ≥ 2 toxicities (according to NCI-CTCAE v5.0). Toxicities must be resolved for at least 2 weeks to Grade 1 or less
4. Patients who have received any prior treatment with compounds targeting PD1, PDL1, CTLA-4, or similar compounds
5. Patients who have previously received trifluridine/tipiracil (TAS-102) or regorafenib
6. Patients with prior exposure to EO2401, EO2040, or EO4010, i.e. therapeutic vaccine compounds including all or some components of EO4010
7. Patients with the following abnormal laboratory values:

   1. Lymphocyte count decreased, grade 2 (lymphocytes <800 - 500/mm3; <0.8 - 0.5 x 109/L), or worse grade
   2. Hemoglobin < 10 g/dL (6.2 mmol/L); transfusion is acceptable to reach the value
   3. Absolute neutrophil count decrease (<1.5 x109/L)
   4. Platelet count decrease (< 75 ×109/L)
   5. Total bilirubin > 1.5 ×upper limit of normal
   6. Alanine aminotransferase (ALT) > 3 ×ULN; if disease metastatic to the liver > 5 xULN
   7. Aspartate aminotransferase (AST) > 3 ×ULN; if disease metastatic to the liver > 5 xULN
   8. Serum creatinine increase (> 1.5 ×ULN)
   9. Abnormal thyroid function per local laboratory levels
8. Other malignancy or prior malignancy with a disease-free interval of less than 3 years prior to ICF signing; except those treated with surgical intervention and an expected low likelihood of recurrence
9. Patients with clinically significant active infection, cardiac disease, significant medical or psychiatric disease/condition
10. Patients with suspected autoimmune or active autoimmune disorder or known history of an autoimmune neurologic condition (e.g., Guillain-Barré syndrome)
11. Patients with a history of solid organ transplantation or allogeneic hematopoietic stem cell transplantation
12. Patients with a history or known presence of tuberculosis
13. Pregnant and breastfeeding patients
14. Patients with a history or presence of human immunodeficiency virus (HIV) and/or active hepatitis B virus (HBV)/hepatitis C virus (HCV)
15. Uncontrolled central nervous system (CNS) metastasis
16. Patients who have received live or attenuated vaccine therapy used for prevention of infectious diseases including seasonal (influenza) vaccinations within 4 weeks of the first dose of study drug
17. Patients with a history of hypersensitivity to any excipient, or active substance, present in the pharmaceutical forms of applicable study treatments
18. Patients under treatment with immunostimulatory or immunosuppressive medications
19. Patients who have received treatment with any other investigational agent, or participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of EO4010 in combination with nivolumab and/or bevacizumab | 12months
  Incidences of AEs, treatment-emergent AEs (TEAEs), Serious Adverse Events (SAEs), deaths, and laboratory abnormalities using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0.

SECONDARY OUTCOMES:
Percentage of patients with shown immunogenicity | 12 months
  Immunogenicity will be assessed by Interferon-γ ELISpot
Overall response rate | 12 months
  Defined as the percentage of patients who have a partial or complete response following Response Evaluation Criteria in Solid Tumors criteria
Disease control rate | 12 months
  Defined as the percentage of patients who have achieved complete response, partial response or stable disease following Response Evaluation Criteria in Solid Tumors criteria
Time to response | 12 months
  Defined as the time interval from first study treatment administration to partial or complete response following Response Evaluation Criteria in Solid Tumors criteria
Duration of response | 12 months
  Defined as the time interval from first study treatment administration to disease progression or death in patients who achieve complete or partial response following Response Evaluation Criteria in Solid Tumors criteria
Progression free survival | 4months
  Defined as the time interval from the date of first study treatment administration to the date of progression following Response Evaluation Criteria in Solid Tumors criteria
Overall survival to the date of death due to any cause. Patients alive will be censored at the date of the last documented follow-up | 12 months
  Defined as the time interval from the date of first study treatment administration to the date of death due to any cause. Patients alive will be censored at the date of the last documented follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fagerberg, Study Director — Enterome
Locations (6):
- MD Anderson, Houston, Texas, United States
- France (3):
  - Hôpital Jean Minjoz, Besançon
  - ICM Val d'Aurelle, Montpellier
  - Saint Antoine hospital, Paris
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Llavero-Hospital Clínico Universitario, Valencia

IPD SHARING:
Plan to Share IPD: No